CLINICAL TRIAL: NCT07000487
Title: Effect of Yoga Training on Nausea and Pain Symptoms in Young Women With Primary Dysmenorrhea: A Randomized Controlled Trial.
Brief Title: Effect of Yoga Training on Nausea and Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Sakine Yılmaz, Assistant Professor Doctor, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Primary dysmenorrhea
Record Dates: First submitted 2025-05-24; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Primary Dysmenorrhea (PD); Yoga
Keywords: primary dysmenorrhea; yoga; pain; nausea; young woman
MeSH Terms: conditions — Pain; Nausea | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: The study consists of two groups: control and experimental group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Since the application will be performed by the researcher, patients will be blinded in this study. The statistician will be blinded in the evaluation of the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental:Yoga (Experimental): Hatha yoga will be applied in this study. Yoga practice will be carried out by the researcher for 6 weeks, 1 day face-to-face and 1 day online, and each practice will be 60 minutes, in total 12 sessions, considering the studies done. It will be applied by a researcher with a yoga certificate. Pre-test and post-test nausea and pain measurements will be made.
  Interventions: Behavioral: Yoga
- No Intervention: Control Group (No Intervention): No application will be made to this group by the researcher.

INTERVENTIONS:
Behavioral: Yoga — Hatha yoga will be applied in this study. Yoga practice will be carried out by the researcher for 6 weeks, 1 day face-to-face and 1 day online, and each practice will be 60 minutes, in total 12 sessions, considering the studies done. It will be applied by a researcher with a yoga certificate. Pre-test and post-test nausea and pain measurements will be made.
  Arms: Experimental:Yoga

SUMMARY:
This study was planned to determine the effect of yoga training on reducing nausea and pain symptoms in young women with primary dysmenorrhea. As a result of this study, evaluating the extent to which women with dysmenorrhea experience pain and nausea and the extent to which yoga has a positive effect on these symptoms may shed light on women experiencing these symptoms and developments in the literature, and may increase the use of non-pharmacological approaches. The results of the study will contribute to the literature on dysmenorrhea, one of the important gynecological problems in women. In addition, although there are many results in the literature on the effectiveness of yoga in the management of nausea symptoms with cancer patients, there are not many studies on nausea on dysmenorrhea. In this respect, it will provide important evidence to the literature.

DETAILED DESCRIPTION:
Primary dysmenorrhea (PD) is one of the most common gynecological conditions affecting an estimated 67% to 90% of young women and is a painful uterine contraction caused by endometrial laceration . PD is also known as painful periods or menstrual cramps that cause pain during the menstrual cycle. Menstrual pain is the most common symptom associated with primary dysmenorrhea. The pathogenesis of menstrual pain is thought to be due to an abnormal increase in the production of vasoactive prostaglandins in the endometrium, which can induce myometrial hyperactivity, uterine tissue ischemia, and pain. The pain caused by dysmenorrhea begins a few days before menstruation and lasts for 48-72 hours. The pain is usually in the pelvis or lower abdomen and may radiate to the lower back and upper thighs. Other symptoms that the individual may experience include diarrhea, headache, stress, and nausea.

Yoga is one of the self-development and exercise methods that fully trains the soul, mind and body and allows the individual to know themselves. Yoga, which is a mental journey that the individual makes to their inner world, is a technique that allows the person to be alone with themselves as a result of the combination of physical posture, breathing techniques and mental meditation. The yoga-based lifestyle includes positive behavioral changes (yamas and niyamas), physical posture practices (asanas), breathing regulation (pranayama), control of the senses (pratyahara) and meditation techniques (dharana, dhyana and samadhi). It has been determined in the literature that yoga reduces menstrual cramps and distress, and it has been reported that it can be used in menstrual problems due to its safety, lack of side effects, low cost, easy accessibility and noninvasiveness. Previous studies report that yoga suppresses menstrual pain by reducing the level of prostaglandin production and myometrial ischemia through "down-regulation of the hypothalamic-pituitary-adrenal axis and the sympathetic nervous system" and has positive effects on psychological well-being. In addition, studies have determined that yoga is also effective in nausea and vomiting symptoms. In a systematic review conducted on individuals with cancer, it was determined that yoga is effective in symptom management (nausea and vomiting, fatigue, anxiety, depression, etc.). The aim of this study is to determine the effect of yoga training in reducing nausea and pain symptoms in young women with primary dysmenorrhea. The results of the study will contribute to the literature on dysmenorrhea, one of the important gynecological problems in women. In addition, although there are many results in the literature on the effectiveness of yoga in the management of nausea and vomiting symptoms with cancer patients, no study on dysmenorrhea has been found. In this respect, it will also provide important evidence to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Having a regular menstrual cycle
* Being single
* Not having any psychiatric diagnosis or gynecological disease (abnormal uterine bleeding, myoma, ovarian cysts, etc.) extremities and any health problems that may prevent physical exercise
* Not having any systemic disease (heart, diabetes, epilepsy, rheumatoid arthritis, etc.)
* Young women who agree to participate in the study and can speak and understand Turkish

Exclusion Criteria:

* Wanting to leave the study, primary dysmenorrhea severity and nausea level below 4 points.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 70 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Before and 6 weeks after yoga practice
  VAS is a suitable measurement tool for the assessment of acute pain. This scale is used to convert some values that cannot be measured numerically. 0 means "No pain" and 10 means "Worst possible pain".
Visual Analog Scale (VAS) | Before and 6 weeks after yoga practice
  VAS will be used to assess nausea.The scale consists of a horizontal line 100 mm/10 cm long. At the left end of the line is 0 "No nausea", while at the right end is 10 "Severe nausea". The individual is asked to mark the point on the line that will accurately reflect their nausea. The distance of the individual's mark to the left end is measured with a ruler. This distance, measured in millimeters, is accepted as a "score" and recorded. In selecting individuals, values of 5 mm and below on the scale are evaluated as "no nausea", and all values of 5 mm and above are evaluated as "experiencing nausea".

CONTACTS AND LOCATIONS:
Locations (1):
- Çankırı, Çankırı, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No